CLINICAL TRIAL: NCT06267235
Title: Dietary Protein, FGF21 and Glucose Homeostasis
Brief Title: Dietary Protein Restriction and Health
Acronym: LOWPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Bente Kiens, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: lowprotein
Record Dates: First submitted 2024-02-07; First posted 2024-02-20 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Protein; Healthy; Diet
Keywords: Protein-restriction; FGF21; Energy; Insulin action

STUDY DESIGN:
Intervention Model Description: Longitudinal study changing diet during the intervention 5 weeks restricted dietary protein + 5 weeks habitual dietary protein consumption
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acute meal test (Experimental): acute intake of a low protein, high carbohydrate diet. No drug intervention
  Interventions: Other: Dietary protein restriction
- Chronic low protein, high carbohydrate diet (Experimental): Low protein, high carbohydrate diet and habitual diet. No drug intervention
  Interventions: Other: Dietary protein restriction
- Low protein , high fat diet (Experimental): Low protein, high fat diet and habitual diet. No drug intervention
  Interventions: Other: Dietary protein restriction

INTERVENTIONS:
Other: Dietary protein restriction — The consumption of different diets restricted in protein replaced by either carbohydrate or fat and an habitual diet.

SUMMARY:
The incidence of type 2 diabetes worldwide has increased significantly over the past decades, which is associated with changing dietary habits and physical inactivity. According to the diet, so far there has been a great focus on the quality of carbohydrates and fat in relation to metabolic health, while the importance of protein has been neglected. The Danes' average protein intake is 1.5 g/kg/day, which is at the high end of the recommendations (0.8-1.5 g/kg/day) from the Nordic Nutrition Recommendations (NNR 2023). Recent studies in rodents have shown that protein restriction has positive effects on health, including improved glucose and insulin homeostasis and reduced fat mass, while a high intake of protein has a negative effect on insulin sensitivity. Previously the investigators have shown, in healthy young men, that consuming a diet low in protein (0.9 g/kg/day), compared to the participants usual diet (1.5 g/kg/day), over 7 days, resulted in an increased insulin sensitivity as well as a marked increase in the plasma fibroblast growth factor 21 (FGF21) concentration. The increased insulin sensitivity is thought to be mediated by the increase in plasma FGF21 concentration. However, the effect is not yet fully understood. It is also not clear whether the increase in plasma FGF21 concentration, as well as the mentioned metabolic effects on insulin and glucose homeostasis, will take place if the participants are kept weight stable on a eucaloric diet.

DETAILED DESCRIPTION:
A three-arm protocol was performed. In protocol 1, participants ingested either a low-protein (LP) meal or a higher protein (HP) meal in a randomized order, separated by 72 h, followed by a 5-week low-protein, high-carbohydrate (LPHC) diet. In protocol 2 and 3, participants ingested either a LPHC diet or a low-protein, high-fat (LPHF) diet for 5 weeks followed by a higher protein diet (HPD) for another 5 weeks. All diets were eucaloric. Resting metabolic rate (RMR) was measured pre, during and post the protein-restricted interventions. A hyperinsulimic-euglycemic clamp was performed post the protein-restricted interventions and post the HPD interventions. A basal subcutaneous abdominal fat biopsy was obtained post the protein-restricted interventions and post the HPD interventions. In a run-in period over 14 days, the participant records the daily number of steps and physical activity, in order to determine their habitual activity level. During this period, a 4-day dietary record is performed, where all ingested food was weighed and recorded. During the experimental period the participant followed the supplied diet. All food consumed during the interventions was handed out to the subject at the institute. All food was packaged and weighed to 1 gram of accuracy. During the dietary intervention, a weekly test in the morning was performed, where the resting metabolic rate was measured and blood samples taken from the arm vein. At week 0, 5 and week 10 body composition was measured by dual energy x-ray absorptiometry scanning (DXA), and the fat biopsy was obtained . At all tests participants arrived fasting at the institute at 8:00 a.m. in the morning. The participant arrived by car or public transport.

ELIGIBILITY:
Inclusion Criteria:

* BMI≤25
* Maximal oxygen uptake ≤42-51 ml/kg/min) • non-smoking

Exclusion Criteria:

* The use of medicine

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Energy balance | from week 0 to week 10.
  Energy balance was measured in an over-night fasted state via indirect calorimetry expressed in MJ/day
  prolonged eucaloric dietary protein restriction compared with a higher habitual protein intake
Insulin sensitivity | Measured at week 5 (low protein, high carbohydrate diet) and week 5 on habitual diet and at week 5 (low protein high fat diet) and week 5 on habitual diet
  Insulin sensitivity was measured by the hyperinsulinemic, euglycemic clamp procedure

SECONDARY OUTCOMES:
Adipose tissue proteomics | After 5 weeks low protein, high carbohydrate and 5 weeks low protein, high fat. On the tenth week on habitual diet
  Mass spectroscopy
Plasma FGF21 | Every week from week 0 to week 10
  Measured by Elisa

CONTACTS AND LOCATIONS:
Overall Officials: Bente Kiens, D.sci, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark